CLINICAL TRIAL: NCT05020912
Title: Alteration of the Immune Microenvironment in Basal Cell Carcinoma (BCC) Following Photodynamic Therapy (PDT)
Brief Title: Alteration of the Immune Microenvironment in Basal Cell Carcinoma Following Photodynamic Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2621
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Aminolevulinic Acid; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: Each participant will serve as their own control - one tumor will be PDT-treated and other left as untreated control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Photodynamic therapy (PDT) (Experimental): Each participant will serve as their own control, receiving PDT for one tumor, no PDT for the second tumor (untreated control).
  Visit 1:
  * Informed consent
  * Blood draw
  * Lesion(s) Photographed
  * (ALA) applied for4 hours
  * PpIX measured in lesions (PpIX buildup monitored every 30 minutes over a 4 h period)
  * PDT with blue light
  Visit 2 (scheduled for within one of the following time intervals: 1-3 days, 4-7 days, or 8-14 days post-PDT):
  * Blood draw
  * Lesion(s) Photographed
  * Mohs surgery
  * After procedure, excess frozen BCC tissue will be saved for analysis
  Interventions: Drug: ALA; Procedure: PDT

INTERVENTIONS:
Drug: ALA — At first visit, ALA applied to one BCC lesion
  Other Names: Levulan
Procedure: PDT — PDT with blue light (for 30 min (~20 mJ/cm2))

SUMMARY:
The purpose of this study is to better understand the immune response to basal cell carcinoma (BCC) treated with Photodynamic Therapy (PDT) in order to develop new methods of treating BCC. Previous research suggests that PDT alters the immune response, possibly in a way that could promote better tumor clearance when combined with other treatments. Overall, participation in this study will help the study team better understand the anti-tumor immune response when BCC is treated with PDT.

DETAILED DESCRIPTION:
PDT is a technique that works by combining a photosensitizing topical agent and an intense light to kill tumor cells. PDT is not currently approved for the treatment of BCC by the Food and Drug Administration (FDA), although it is approved for that purpose in many European countries.

This is an internally (bilaterally) controlled trial that will enroll 24 participants with biopsy-proven BCC who are planning to undergo tumor removal via Mohs surgery. Within this cohort, one tumor will be PDT-treated and the other left as an untreated control. This study is also a cohort-controlled trial, because discarded tissue from fully de-identified Mohs participants will be analyzed after routine Mohs surgery, in order to establish the baseline variability in tumor-infiltrating immune cell parameters in non-PDT-treated participants.

The objectives of this study are:

To determine the time to maximum expression of immune checkpoint molecules in BCC tumors and peri-tumoral stroma after PDT, as compared to untreated tumors.

To determine the ratio of cytotoxic T cells to regulatory T cells in BCC tumors and peri-tumoral stroma after PDT, as compared to untreated tumors.

To determine whether circulating T-cells, collected from patients' peripheral blood, sampled before and after PDT treatment of a BCC tumor, show a higher proportion of tumor-activated CD8+ T-cells after PDT. The hypothesis is that PDT of the localized tumor will trigger a systemic anti-tumor immune effect.

To determine the rate of protoporphyrin IX (PpIX) accumulation and maximal PpIX levels.in tumors To determine the rate of production and maximal levels of singlet oxygen (O2) produced during blue light exposure To assess change in the volume, color, and appearance of tumors at the Mohs surgery visit compared to the PDT visit To assess for distant tumor (abscopal) effects after PDT

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled to undergo Mohs surgery within the Dermatologic Surgery unit of the Department of Dermatology, Cleveland Clinic
* Must have at least one BCC tumor eligible for removal by surgical excision
* Men and women of any ethnic group are eligible
* Must provide informed consent to participate

Exclusion Criteria:

* Pregnant or breastfeeding
* Currently being treated for other cancers with medical or radiation therapy
* Known hypersensitivity to 5-aminolevulinic acid (ALA)
* History of a photosensitivity disease, e.g.,porphyria cutanea tarda

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to maximum expression of immune checkpoint molecules | at visit 2 (1-14 days)
  Time (days) to maximum expression of immune checkpoint molecules in BCC tumors and peri-tumoral stroma after PDT, as compared to untreated tumors.
  Data from frozen BCC specimens post-PDT by immunostaining the tumor specimens with antibodies against PD-L1, PD-1, CTLA-4 as well as the newer IC molecules TIGIT, TIM-3, and LAG-3
Altered expression of immune checkpoint molecules | at visit 2 (1-14 days)
  Altered expression of immune checkpoint molecules in BCC tumor specimens after PDT.
  Assessed by comparing IC molecule expression in PDT treated and untreated tumors with immunostaining in the tumor specimens with antibodies against PD-L1, PD-1, CTLA-4 as well as the newer IC molecules TIGIT, TIM-3, and LAG-3. (quantifying with immunofluorescence microscope)
Altered recruitment of different immune cell subtypes in BCC tumor specimens | at visit 2 (1-14 days)
  Determine the ratio of cytotoxic T cells to regulatory T cells in BCC tumors and peri-tumoral stroma after PDT, as compared to untreated tumors.
  Measured with specific antibodies against the following markers, to determine the qualitative time course of infiltration by each immune cell populations: Neutrophils (Gr1+ or MPO+); Macrophages(F4/80+); MDSCs (CD33, S100A9); cytotoxicT-cells(CD8+); regulatory T-cells(CD4+,FoxP3+,CD25+, CD127-); NK natural killer cells(CD56+CD16+).

SECONDARY OUTCOMES:
Proportion of tumor-activated CD8+ T-cells after PDT | at visit 2 (1-14 days)
  Difference in CD8 T cells after PDT collected from participants' peripheral blood, sampled before and after PDT treatment of a BCC tumor.
  This data is derived from patient blood samples. Each patient will have two blood draws: at Visit 1 (before PDT, to establish a baseline) and at Visit 2. We will compare the proportion of CD8 T cells after PDT based on when the participant returns (within the 3 time ranges), and a single value (difference in CD8 T cells, measured before and after PDT) will be reported for that patient.
Rate of protoporphyrin IX (PpIX) accumulation in tumors | Every 30 minutes up to 4 hours
  Relative rate of PpIX accumulation in tumors assessed via noninvasive measurements of PpIX fluorescence using a dosimeter.
  PpIX will be measured every 30 minutes during the 4 hour incubation. The purpose is to monitor PDT kinetics. We will measure the level of PpIX at each time point, but the final outcome to report is relative rate of change in fluorescence intensity.
Maximal PpIX levels in tumors | Every 30 minutes up to 4 hours
  Maximal PpIX levels in tumors, assessed via noninvasive measurements of PpIX fluorescence using a dosimeter
Change in the color of tumors | at visit 1 (pre PDT) and visit 2 (1-14 days)
  Change in the color of tumors as reported by the participants at the Mohs surgery visit compared to the PDT visit. Number of participants that report common findings after PDT.
Change in the appearance of tumors | at visit 1 (pre PDT) and visit 2 (1-14 days)
  Change in the appearance of tumors as reported by the participants at the Mohs surgery visit compared to the PDT visit. Number of participants that report common findings after PDT. Appearance as being the shape, texture and overlying skin changes.
Change in the volume of tumors | at visit 1 (pre PDT) and visit 2 (1-14 days)
  Change in the volume of tumors at the Mohs surgery visit compared to the PDT visit.
  Tumor volumes (mm3) will be determined from computerized analysis of 3-D photographs.
Distant tumor (abscopal) effects after PDT | at visit 2 (1-14 days)
  Number and type of immune cell present, expression of immune checkpoint molecules, and tumor-activated CD8 T cells present in blood compared to archived samples that did not receive PDT.
To determine the relationship of PDT with the expression of immune- and cancer-associated RNA molecules | at visit 1 (pre PDT) and visit 2 (1-14 days)
  Determine whether PDT is associated with altered expression of immune- and cancer-associated RNA transcripts in BCC using NanoString nCounter.

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Maytin, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, SAP, ICF, CSR